CLINICAL TRIAL: NCT05301582
Title: The Ability of Tidal Volume Challenge Test to Predict Early Post- Operative Acute Kidney Injury and Intra-operative Hypotension in Laparoscopic Abdominal Surgeries. Prospective Observational Study.
Brief Title: T.V Challenge to Predict Early Post- Operative Acute Kidney Injury and Intra-operative Hypotension in Laparoscopic Abdominal Surgeries
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Hala Mostafa Gomaa (Unknown); Ahmed Mohamed Ahmed Mostafa (Unknown); Mohamed Abdel Ghany Ali Elshazly (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Other Study IDs: M.D- 302-2021
Record Dates: First submitted 2022-02-12; First posted 2022-03-29 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Tidel Volume Challenge Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group: A total of 70 consecutive adult patients, aged 18-65 years scheduled for elective laparoscopic surgery under general anesthesia will be included in the study.
  Interventions: Diagnostic Test: Tidal volume challenge test

INTERVENTIONS:
Diagnostic Test: Tidal volume challenge test — The purpose of our study is to verify the predictability of TVC test during laparoscopic abdominal surgery for early postoperative AKI and intra-operative hypotension.

SUMMARY:
The purpose of study is to verify the predictability of TV Chalange test during laparoscopic abdominal surgery for early postoperative AKI and intra-operative hypotension.

.

DETAILED DESCRIPTION:
The number and scope of laparoscopic surgery are increasing. Now almost every abdominal organ seems suitable for laparoscopic surgery. Laparoscopy may be considered potentially risky because it may involve extreme changes in the patient's position, prolonged intra-abdominal insufflation and carbon dioxide (CO2) degassing, unexpected visceral damage, and difficulty in assessing blood loss. The anesthesiologist must select the appropriate anesthesia management technique, conduct proper monitoring, and be aware of potential complications. Early detection and reduction of possible intra-operative problems can prevent postoperative complications and early complications.

Laparoscopic injection of CO2 or N2O can cause cardiovascular depression . Insufflation at a high flow rate can also exacerbate cardiovascular sequelae, including hypotension and bradycardia, and cause cardiac arrest . Intra-operative hypotension caused by rapid laparoscopic inflation is caused by the vagal-mediated cardiovascular reflex caused by the rapid expansion of the peritoneum. It can also be attributed to the reduction in preload and venous return associated with the pneumo-peritoneum (PP) .

During the period of elevated intra-abdominal pressure, there are three different mechanisms of renal insufficiency, including hypercapnia caused by CO2 insufflation, elevated intra-abdominal pressure and renin-angiotensin-aldosterone system (RAAS) .

In another study, the incidence of AKI after laparoscopic abdominal surgery was 35.9%, which was higher than the previous study .

Patients with low-volume status are susceptible to AKI due to ischemic acute tubular necrosis due to renal insufficiency, and predisposed by hypotension as a pre-renal cause.

Although low volume status has a major role in post-operative AKI .Yet, there are rising theories explaining the increased incidence of AKI in patients undergoing laparoscopic surgeries to increased renal resistive index (RRI) by increased intra-abdominal pressure Intra-operative volume status indicators are variable, including inferior vena cava (IVC), carotid artery ratio (JCR), stroke volume change (SVV) and pulse pressure change (PPV). These indicators may be reliable, but complex, time-consuming, and require trained personnel and high-tech equipment .

The Tidal Volume Challenge (TVC) test is a new tool which is used to assess the volume status and it has been approved as a reliable tool in neurosurgery patients . However, as far as we know, it has not been used to predict hypotension and AKI in laparoscopic surgeries. We hypothesis that mimicking the effect of increased intra-abdominal pressure transiently for a short period of time by TVC test could contribute in detecting patients at high risk of developing post-operative AKI.

TVC test/ abdominal insufflation adverse consequences can be also explained mainly by reduced venous compliance in some patients leading to mobilization of blood to peripheral venous system, with reduced venous elasticity the passive blood recoil to the heart maintaining hemo-dynamic stability and organ perfusion will be diminished, aggravating the effect of increased intra-abdominal or intra-thoracic pressure. That mechanism has been studied in orthostatic hypotension The purpose of study is to verify the predictability of TVC test during laparoscopic abdominal surgery for early postoperative AKI and intra-operative hypotension.

.

ELIGIBILITY:
Inclusion Criteria:

* Gender both males and females
* ASA Class I and II
* Age 18-65 years
* Patients undergoing elective laparoscopic surgery under general anaesthesia

Exclusion Criteria:

* Kidney dysfunction
* Cardiac arrhythmias and valvular heart disease
* Chronic obstructive pulmonary disease
* Right ventricular failure
* Intracranial hypertension
* Airway asthma or a long history of smoking
* Those who are on NSAID for 1 week prior to surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in Kasr Alainy Hospital of Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
The sensitivity of TVC test to predict early post-operative AKI in laparoscopic surgeries. | Through Study Completionan average of 24 hours
  The sensitivity of TVC test to predict early post-operative AKI in laparoscopic surgeries.

SECONDARY OUTCOMES:
The sensitivity of TVC test to predict intraoperative post insufflation and desufflation hypotension. | Through Study Completionan average of 24 hours
  The sensitivity of TVC test to predict intraoperative post insufflation and desufflation hypotension.
The relationship between exposure index (the product of inflation time x intra-abdominal pressure) and early post-operative AKI. | Through Study Completionan average of 24 hours
  The relationship between exposure index (the product of inflation time x intra-abdominal
The incidence of AKI in laparoscopic surgeries. | Through Study Completionan average of 24 hours
  The incidence of AKI in laparoscopic surgeries.
The ability of (uNGAL) to predict early post operative AKI. | Through Study Completionan average of 24 hours
  The ability of (uNGAL) to predict early post operative AKI.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Mohamed, M.D, Principal Investigator — Cairo University; Hala M Gomaa, M.D, Principal Investigator — Cairo University; Mohamed A Ali Elshazly, M.D, Study Director — Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided